CLINICAL TRIAL: NCT05450367
Title: Predictive Markers of Response and Toxicity in Patients With a Haematological Malignancy Treated With Immunotherapy.
Acronym: PRONOSTIM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220632
Record Dates: First submitted 2022-06-27; First posted 2022-07-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Blood Cancer
Keywords: Haematologic malignancies; Immunotherapy; Response predictor; Immune-related adverse event
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with a haematological malignancy treated with immunotherapy
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection

SUMMARY:
Immunotherapies have substantially improved the prognosis of patients with haematological malignancies. While clinical trial data suggest durable complete response rates, markers associated with non-response to treatment are still poorly described. The identification of predictive markers using demographic, physiologic, biologic, immunologic data as well as patients' treatment history, might enable the optimization of therapeutic sequences and the reduction of treatment toxicity.

This study aim to assess markers of toxicity and response following an immunotherapy in patients with a haematological malignancy using real life data.

It will allow the development of clinical and therapeutic benchmarks to guide medical decisions in relation to the therapeutic strategies to be implemented for patients benefiting from real-life conditions, in addition to the results obtained in randomized studies.

ELIGIBILITY:
Inclusion Criteria :

* adult >or= 18 years old,
* Suffering from one of the following pathologies: Hodgkin's lymphoma, Diffuse large B-cell lymphoma, Mantle B-cell lymphoma, Acute myeloid leukemia, Acute lymphoid leukemia, Peripheral T-cell lymphoma,
* Patients treated wuth any of the following immunotherapy : nivolumab, pembrolizumab, brentuximab vedotin, axicabtagene ciloleucel, tisagenlecleucel, brexucabtagene autoleucel, gentuzumab ozogamicine, polatuzumab vedotin and blinatumomab,

Exclusion Criteria :

- Patients opposed to the collection of their personnal data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with a haematological malignancy and treated with immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Proportion of complete response | Through study completion, an average of 1 year
  Treatment response : Explore the proportion of complete response
Proportion of partial response | Through study completion, an average of 1 year
  Treatment response : Explore the proportion of partial response
Proportion of stable disease | Through study completion, an average of 1 year
  Treatment response : Explore the proportion of stable disease
Proportion of progress disease | Through study completion, an average of 1 year
  Treatment response : Explore the proportion of progress disease

SECONDARY OUTCOMES:
Incidence of grade III adverse events | Through study completion, an average of 1 year
  Toxicity : Explore the cumulative incidence of grade III and IV adverse events
Incidence of grade IV adverse events | Through study completion, an average of 1 year
  Toxicity : Explore the cumulative incidence of grade III and IV adverse events
Interruption rates of immunotherapy | Through study completion, an average of 1 year
  Toxicity : Explore the interruption and discontinuation rates of immunotherapy
Discontinuation rates of immunotherapy | Through study completion, an average of 1 year
  Toxicity : Explore the interruption and discontinuation rates of immunotherapy
Time interval between the date of initiation treatment and the date of first progression | Through study completion, an average of 1 year
  Progression free survival
Time interval between the date of initiation treatment and the date of death from any cause | Through study completion, an average of 1 year
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Zerbit, PharmD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique - Hôpitaux de Paris (AP-HP) - Cochin Hospital, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Detroit M, Collier M, Beeker N, Willems L, Decroocq J, Deau-Fischer B, Vignon M, Birsen R, Moufle F, Leclaire C, Balladur E, Deschamps P, Chauchet A, Batista R, Limat S, Treluyer JM, Ricard L, Stocker N, Hermine O, Choquet S, Morel V, Metz C, Bouscary D, Kroemer M, Zerbit J. Predictive Factors of Response to Immunotherapy in Lymphomas: A Multicentre Clinical Data Warehouse Study (PRONOSTIM). Cancers (Basel). 2023 Aug 9;15(16):4028. doi: 10.3390/cancers15164028. PMID 37627056